CLINICAL TRIAL: NCT02320721
Title: A Randomized, Open-label, 2-arm Parallel-group, Multicenter, 26-week Study Assessing the Safety and Efficacy of H0E901-U300 Versus Lantus in Older Patients With Type 2 Diabetes Inadequately Controlled on Antidiabetic Regimens Either Including no Insulin, or With Basal Insulin as Their Only Insulin
Brief Title: Comparison of the Safety and Efficacy of HOE901-U300 With Lantus in Older Patients With Type2 Diabetes Insufficiently Controlled on Their Current Antidiabetic Medications
Acronym: SENIOR
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC13799; 2014-002399-10; U1111-1159-3018 (Other: UTN)
Record Dates: First submitted 2014-12-16; First posted 2014-12-19 (Estimated); Results first posted 2017-07-11 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- HOE901-U300 (Experimental): HOE901-U300 (Insulin glargine, 300 U/mL) once daily up to Week 26 on top of stable non-insulin antihyperglycemic therapy.
  Interventions: Drug: Insulin Glargine (HOE901 - U300); Drug: Background therapy
- Lantus (Active Comparator): Lantus (Insulin glargine, 100 U/mL) once daily up to Week 26 on top of stable non-insulin antihyperglycemic therapy.
  Interventions: Drug: Insulin Glargine (HOE901 - U100); Drug: Background therapy

INTERVENTIONS:
Drug: Insulin Glargine (HOE901 - U300) — Self-administered by subcutaneous (SC) injection in the evening using a pre-filled pen. Dose titration to achieve fasting self-monitored plasma glucose (SMPG) from 90 to 130 mg/dL (5.0 to 7.2 mmol/L).
  Other Names: Toujeo®
  Arms: HOE901-U300
Drug: Insulin Glargine (HOE901 - U100) — Self-administered by SC injection in the evening using a pre-filled pen. Dose titration to achieve fasting SMPG from 90 to 130 mg/dL (5.0 to 7.2 mmol/L).
  Other Names: Lantus®
  Arms: Lantus
Drug: Background therapy — Non-insulin anti-diabetic drugs with the exception of thiazolidinediones.

SUMMARY:
Primary Objective:

To demonstrate the non-inferiority of H0E901-U300 to Lantus, in change of glycated hemoglobin A1c (HbA1c).

Secondary Objectives:

To demonstrate the superiority of H0E901-U300 in comparison with Lantus in:

* Percentage of participants with at least one severe and/or confirmed (by plasma glucose ≤70mg/dL [3.9mmol/L]) hypoglycemia event from 22:00 to 08:59 next morning
* Percentage of participants with at least one nocturnal (from 00:00-05:59) severe and/or confirmed (≤70mg/dL [3.9mmol/L]) hypoglycemia event
* Percentage of participants with at least one severe and/or confirmed (by plasma glucose ≤70mg/dL [3.9mmol/L]) hypoglycemia event occurring at any time of day
* HbA1c change

DETAILED DESCRIPTION:
The study consisted of a 4-week screening period, a 26-week treatment period comparing HOE901-U300 to Lantus, and a 2-day safety follow-up period.

ELIGIBILITY:
Inclusion criteria:

* Participants ≥65 years old with type 2 diabetes mellitus, inadequately controlled on antidiabetic regimens either including no insulin, or with basal insulin as their only insulin.
* Signed informed consent.

Exclusion criteria:

* HbA1c at screening visit:

  * <7.0% or >10.0% for participants taking basal insulin.
  * <7.5% or >11.0% for insulin-naïve participants.
* History of type 2 diabetes mellitus for less than 1 year before screening.
* Participants not on stable basal insulin dose (±10% in the last 8 weeks prior to screening visit).
* Change in dose of antidiabetic treatment or initiation of new glucose-lowering medications in the last 8 weeks prior to screening.
* Chronic (>10 days continuous use in previous 6 months) use of bolus insulin injections, whether given separately or as part of a combination with basal insulin, e.g. premix insulin; For insulin-naïve individuals: current or previous insulin use except for a maximum of 10 consecutive days (e.g. acute illness, surgery) during the last year prior to screening.
* Cognitive disorder and dementia assessed clinically and by Mini-Mental State Examination (MMSE) score <24, or any neurologic disorder that would likely affect the participant's ability to follow the study procedure. The participant would be eligible despite an MMSE score <24 if the investigator determined that the low score reflected educational or cultural background and not dementia as long as the participant was otherwise able to meet the study requirements.
* Participants who had end-stage renal disease (<15 mL/min/1.73m^2, per estimated Glomerular filtration rate (eGFR) measurement by Modification of Diet in Renal Disease (MDRD).

The above information was not intended to contain all considerations relevant to a participant's potential participation in a clinical trial.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1014 (Actual)
Dates: Start 2015-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (162):
- United States (64):
  - Investigational Site Number 840058, Saraland, Alabama
  - Investigational Site Number 840019, Fresno, California
  - Investigational Site Number 840021, Fresno, California
  - Investigational Site Number 840040, Greenbrae, California
  - Investigational Site Number 840070, Huntington Park, California
  - Investigational Site Number 840064, Los Angeles, California
  - Investigational Site Number 840031, Norwalk, California
  - Investigational Site Number 840065, Oakland, California
  - Investigational Site Number 840050, Orange, California
  - Investigational Site Number 840036, Simi Valley, California
  - Investigational Site Number 840003, Temecula, California
  - Investigational Site Number 840062, Walnut Creek, California
  - Investigational Site Number 840027, Longmont, Colorado
  - Investigational Site Number 840030, Bradenton, Florida
  - Investigational Site Number 840010, Miami, Florida
  - Investigational Site Number 840035, Miami, Florida
  - Investigational Site Number 840014, New Port Richey, Florida
  - Investigational Site Number 840051, Ocoee, Florida
  - Investigational Site Number 840056, Palm Harbor, Florida
  - Investigational Site Number 840007, St. Petersburg, Florida
  - Investigational Site Number 840041, Roswell, Georgia
  - Investigational Site Number 840053, Statesboro, Georgia
  - Investigational Site Number 840042, Woodstock, Georgia
  - Investigational Site Number 840005, Arlington Heights, Illinois
  - Investigational Site Number 840004, Peoria, Illinois
  - Investigational Site Number 840029, Springfield, Illinois
  - Investigational Site Number 840013, Avon, Indiana
  - Investigational Site Number 840023, Avon, Indiana
  - Investigational Site Number 840039, Evansville, Indiana
  - Investigational Site Number 840006, Muncie, Indiana
  - Investigational Site Number 840026, Des Moines, Iowa
  - Investigational Site Number 840033, West Des Moines, Iowa
  - Investigational Site Number 840032, Overland Park, Kansas
  - Investigational Site Number 840069, Metairie, Louisiana
  - Investigational Site Number 840020, Flint, Michigan
  - Investigational Site Number 840037, Nashua, New Hampshire
  - Investigational Site Number 840018, New York, New York
  - Investigational Site Number 840048, Asheville, North Carolina
  - Investigational Site Number 840009, Charlotte, North Carolina
  - Investigational Site Number 840011, Greensboro, North Carolina
  - Investigational Site Number 840047, Greenville, North Carolina
  - Investigational Site Number 840016, Salisbury, North Carolina
  - Investigational Site Number 840012, Wilmington, North Carolina
  - Investigational Site Number 840022, Fargo, North Dakota
  - Investigational Site Number 840072, Cincinnati, Ohio
  - Investigational Site Number 840054, Wadsworth, Ohio
  - Investigational Site Number 840067, Bend, Oregon
  - Investigational Site Number 840057, Corvallis, Oregon
  - Investigational Site Number 840045, Feasterville, Pennsylvania
  - Investigational Site Number 840017, Pittsburgh, Pennsylvania
  - Investigational Site Number 840059, Greenville, South Carolina
  - Investigational Site Number 840015, Greer, South Carolina
  - Investigational Site Number 840002, Chattanooga, Tennessee
  - Investigational Site Number 840046, Chattanooga, Tennessee
  - Investigational Site Number 840034, Knoxville, Tennessee
  - Investigational Site Number 840055, Arlington, Texas
  - Investigational Site Number 840001, Dallas, Texas
  - Investigational Site Number 840024, Irving, Texas
  - Investigational Site Number 840061, North Richland Hills, Texas
  - Investigational Site Number 840028, Richmond, Texas
  - Investigational Site Number 840063, San Antonio, Texas
  - Investigational Site Number 840038, St. George, Utah
  - Investigational Site Number 840025, Federal Way, Washington
  - Investigational Site Number 840060, Bridgeport, West Virginia
- Argentina (5):
  - Investigational Site Number 032001, Caba
  - Investigational Site Number 032002, Caba
  - Investigational Site Number 032006, Capital Federal
  - Investigational Site Number 032004, Ciudad Autonoma de Buenos Aire
  - Investigational Site Number 032003, Mar del Plata
- Australia (4):
  - Investigational Site Number 036002, Box Hill
  - Investigational Site Number 036004, Fitzroy
  - Investigational Site Number 036001, Geelong
  - Investigational Site Number 036003, Herston
- Canada (10):
  - Investigational Site Number 124003, Brampton
  - Investigational Site Number 124005, Burlington
  - Investigational Site Number 124008, Chatham
  - Investigational Site Number 124010, Mirabel
  - Investigational Site Number 124009, Montreal
  - Investigational Site Number 124006, Sainte-Foy
  - Investigational Site Number 124004, Thornhill
  - Investigational Site Number 124002, Toronto
  - Investigational Site Number 124001, Vancouver
  - Investigational Site Number 124007, Vancouver
- Colombia (5):
  - Investigational Site Number 170004, Armenia
  - Investigational Site Number 170007, Barranquilla
  - Investigational Site Number 170001, Bogotá
  - Investigational Site Number 170005, Bogotá
  - Investigational Site Number 170003, Manizales
- France (3):
  - Investigational Site Number 250004, Lyon
  - Investigational Site Number 250006, Nantes
  - Investigational Site Number 250005, Poitiers
- Germany (5):
  - Investigational Site Number 276004, Dresden
  - Investigational Site Number 276003, Essen
  - Investigational Site Number 276001, München
  - Investigational Site Number 276005, Potsdam
  - Investigational Site Number 276002, Saarlouis
- Hungary (8):
  - Investigational Site Number 348004, Balatonfüred
  - Investigational Site Number 348001, Budapest
  - Investigational Site Number 348005, Budapest
  - Investigational Site Number 348007, Budapest
  - Investigational Site Number 348003, Budapest
  - Investigational Site Number 348008, Csongrád
  - Investigational Site Number 348009, Debrecen
  - Investigational Site Number 348002, Gyula
- Italy (5):
  - Investigational Site Number 380004, Bologna
  - Investigational Site Number 380005, Chieti
  - Investigational Site Number 380003, Genova
  - Investigational Site Number 380002, Milan
  - Investigational Site Number 380001, Milan
- Japan (7):
  - Investigational Site Number 392008, Adachi-Ku
  - Investigational Site Number 392003, Atsugi-Shi
  - Investigational Site Number 392002, Kamakura-Shi
  - Investigational Site Number 392010, Sagamihara-Shi
  - Investigational Site Number 392004, Sakado-Shi
  - Investigational Site Number 392013, Sapporo
  - Investigational Site Number 392012, Sendai
- Mexico (4):
  - Investigational Site Number 484002, Aguascalientes
  - Investigational Site Number 484004, Cuernavaca
  - Investigational Site Number 484001, Guadalajara
  - Investigational Site Number 484003, Monterrey
- Peru (7):
  - Investigational Site Number 604004, Arequipa
  - Investigational Site Number 604007, Ica
  - Investigational Site Number 604002, Lima
  - Investigational Site Number 604005, Lima
  - Investigational Site Number 604001, Lima
  - Investigational Site Number 604006, Lima
  - Investigational Site Number 604003, Piura
- Poland (5):
  - Investigational Site Number 616005, Lublin
  - Investigational Site Number 616004, Szczecin
  - Investigational Site Number 616003, Warsaw
  - Investigational Site Number 616002, Warsaw
  - Investigational Site Number 616001, Zabrze
- Romania (7):
  - Investigational Site Number 642006, Bacau
  - Investigational Site Number 642001, Bucharest
  - Investigational Site Number 642007, Constanța
  - Investigational Site Number 642004, Oradea
  - Investigational Site Number 642005, Sibiu
  - Investigational Site Number 642002, Târgu Mureş
  - Investigational Site Number 642003, Târgu Mureş
- South Korea (5):
  - Investigational Site Number 410003, Seoul
  - Investigational Site Number 410005, Seoul
  - Investigational Site Number 410002, Seoul
  - Investigational Site Number 410001, Seoul
  - Investigational Site Number 410004, Wŏnju
- Spain (8):
  - Investigational Site Number 724008, A Coruña
  - Investigational Site Number 724004, Alzira
  - Investigational Site Number 724001, Badalona
  - Investigational Site Number 724002, Ferrol
  - Investigational Site Number 724006, Málaga
  - Investigational Site Number 724007, Quart de Poblet
  - Investigational Site Number 724003, Sanlúcar de Barrameda
  - Investigational Site Number 724005, Seville
- Sweden (4):
  - Investigational Site Number 752002, Gothenburg
  - Investigational Site Number 752004, Härnösand
  - Investigational Site Number 752003, Rättvik
  - Investigational Site Number 752001, Västra Frölunda
- United Kingdom (6):
  - Investigational Site Number 826003, Belfast
  - Investigational Site Number 826005, Belfast
  - Investigational Site Number 826001, Bristol
  - Investigational Site Number 826004, Redhill
  - Investigational Site Number 826006, Rotherham
  - Investigational Site Number 826002, Swansea

REFERENCES:
- [Result] Ritzel R, Harris SB, Baron H, Florez H, Roussel R, Espinasse M, Muehlen-Bartmer I, Zhang N, Bertolini M, Brulle-Wohlhueter C, Munshi M, Bolli GB. A Randomized Controlled Trial Comparing Efficacy and Safety of Insulin Glargine 300 Units/mL Versus 100 Units/mL in Older People With Type 2 Diabetes: Results From the SENIOR Study. Diabetes Care. 2018 Aug;41(8):1672-1680. doi: 10.2337/dc18-0168. Epub 2018 Jun 12. PMID 29895556

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 162 study centers across 18 countries. A total of 1515 participants were screened between 16 January 2015 and 14 October 2015, of whom 501 were screen failures.
Pre-assignment Details: A total of 1014 participants were randomized in 1:1 ratio to either HOE901-U300 or Lantus, stratified by screening hemoglobin A1c (HbA1c) values (<8% or ≥8%); previous use of insulin (insulin-naïve versus pre-treated); and use of sulfonylurea or meglitinides at screening ('yes' versus 'no').
Groups:
- HOE901-U300: HOE901-U300 (Insulin glargine, 300 U/mL) subcutaneous (SC) injection once daily up to Week 26 on top of stable non-insulin antihyperglycemic therapy.
- Lantus: Lantus (Insulin glargine, 100 U/mL) SC injection once daily up to Week 26 on top of stable non-insulin antihyperglycemic therapy.
Period: Overall Study
Arm/Group | HOE901-U300 | Lantus
Started | 508 | 506
Treated (Safety Population) | 508 | 505
Completed | 481 | 472
Not Completed | 27 | 34
Not completed — Adverse Event | 6 | 6
Not completed — Lack of Efficacy | 2 | 0
Not completed — Poor compliance to protocol | 3 | 7
Not completed — Randomized but not treated | 0 | 1
Not completed — Hypoglycemia | 1 | 0
Not completed — Other than specified above | 15 | 20

BASELINE CHARACTERISTICS:
Population: Baseline population included all randomized participants.
Groups:
- HOE901-U300: HOE901-U300 (Insulin glargine, 300 U/mL) SC injection once daily up to Week 26 on top of stable non-insulin antihyperglycemic therapy.
- Total: Total of all reporting groups
Arm/Group | HOE901-U300 | Lantus | Total
Number analyzed (Participants) | 508 | 506 | 1014
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.1 (4.9) | 70.8 (4.8) | 71.0 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 258 | 229 | 487
  Male | 250 | 277 | 527
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — Population: Number of participants analyzed = participants with available data for this baseline measure.
  kg/m^2
    number analyzed (Participants) | 508 | 505 | 1013
    (all) | 30.9 (5.5) | 31.2 (5.7) | 31.1 (5.6)
Duration of Type 2 Diabetes [Mean (Standard Deviation); unit: years] | 15.29 (8.17) | 15.35 (7.70) | 15.32 (7.93)
Baseline Glycated Hemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: percentage of HbA1c] | 8.20 (0.91) | 8.22 (0.92) | 8.21 (0.91)
Randomization strata of insulin [Count of Participants; unit: Participants]
  Insulin-naive | 166 | 165 | 331
  Insulin pre-treated | 342 | 341 | 683
Age Group [Count of Participants; unit: Participants]
  <75 years of age | 373 | 400 | 773
  ≥75 years of age | 135 | 106 | 241

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline to Week 26
Description: Adjusted least square (LS) means were obtained from analysis of covariance (ANCOVA) after multiple imputation of missing data including post baseline HbA1c data during the 26-week randomized period.
Time Frame: Baseline, Week 26
Population: Intent-to-treat (ITT) population included all randomized participants regardless of whether the treatment kit was used, and analyzed according to the treatment group allocated by randomization.
Measure: Least Squares Mean (Standard Error); unit: percentage of hemoglobin
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 506
percentage of hemoglobin | -0.89 (0.038) | -0.91 (0.042)
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Analysis was performed using ANCOVA model including the fixed categorical effects of treatment group, randomization strata, as well as the continuous fixed covariates of baseline value and following multiple imputation procedure for missing data; Test type: Non-Inferiority — Non-inferiority of HOE901-U300 vs Lantus was demonstrated if the upper bound of the two-sided 95% confidence interval (CI) for the difference between groups was <0.3%; LS Mean Difference = 0.02, 95% CI 2-sided [-0.092 to 0.129], Standard Error of Mean 0.056

2. Secondary Outcome: Percentage of Participants With At Least One Severe and/ or Confirmed (≤3.9 mmol/L [70 mg/dL]) Nocturnal Hypoglycemia (22:00 to 08:59 Hours Next Morning) During 26-Week Randomized Period
Description: Estimated percentages from multiple imputation approach including data from the 26-week randomized period. Severe hypoglycemia was an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Confirmed hypoglycemia was an event associated with plasma glucose ≤3.9 mmol/L (70 mg/dL).
Time Frame: Baseline up to Week 26
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 506
percentage of participants | 48.3 | 47.7
Statistical Analysis 1: Comparison: HOE901-U300 vs Lantus; Analysis was done by Cochran-Mantel-Haenszel method with randomization strata (screening HbA1c [<8.0%; ≥8.0%], previous use of insulin [naive, pre-treated], use of sulfonylurea or meglitinides at screening [yes, no]), following multiple imputation procedure for missing data; Test type: Superiority or Other — A hierarchical testing procedure was used to control type I error and handle multiple endpoint analyses. Testing was then performed sequentially in the order the endpoints are reported. The hierarchical testing sequence continued only if previous endpoint was statistically significant at 0.05 level; p = 0.8415, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level; Relative risk = 1.01, 95% CI 2-sided [0.890 to 1.153]

3. Secondary Outcome: Percentage of Participants With At Least One Severe and/ or Confirmed (≤3.9 mmol/L [70 mg/dL]) Nocturnal Hypoglycemia (00:00 to 05:59 Hours) During 26-Week Randomized Period
Description: as for outcome 2
Time Frame: Baseline up to Week 26
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 506
percentage of participants | 20.2 | 22.5

4. Secondary Outcome: Percentage of Participants With At Least One Severe and/ or Confirmed (≤3.9 mmol/L [70 mg/dL]) Hypoglycemia Occurring at Any Time of the Day During 26-Week Randomized Period
Description: as for outcome 2
Time Frame: Baseline up to Week 26
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 506
percentage of participants | 59.4 | 62.7

5. Secondary Outcome: Percentage of Participants With HbA1c <7.5% or HbA1c <7% During 26-Week Randomized Period
Description: Participants without any available HbA1c assessment at Week 26 were considered as non-responders in the analyses.
Time Frame: Baseline up to Week 26
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 506
percentage of participants
  HbA1c <7.5% | 60.6 | 58.9
  HbA1c <7.0% | 33.3 | 35.2

6. Secondary Outcome: Percentage of Participants With HbA1c <7.5% or <7.0% at Week 26 and No Severe and/or Confirmed (≤3.9 mmol/L [70 mg/dL]) Hypoglycemia During 26-Week Randomized Period
Description: Severe hypoglycemia was an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions. Confirmed hypoglycemia was an event associated with plasma glucose ≤3.9 mmol/L (70 mg/dL).
Time Frame: Baseline up to Week 26
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 506
percentage of participants
  HbA1c <7.5% | 26.4 | 21.5
  HbA1c <7.0% | 14.0 | 12.3

7. Secondary Outcome: Change in Fasting Plasma Glucose (FPG) From Baseline to Week 26
Description: Adjusted LS means from multiple imputation approach including post baseline values during the 26-week randomized period.
Time Frame: Baseline, Week 26
Population: ITT population. Here 'Overall number of participants analyzed' signifies participants with available data for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: mmol/L
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 484 | 482
mmol/L | -1.68 (0.122) | -1.77 (0.135)

8. Secondary Outcome: Change in World Health Organization-5 (WHO-5) Well-Being Questionnaire Percentage Score From Baseline to Week 26
Description: WHO-5 well-being index evaluates positive psychological well-being during the past 2 weeks and consists of 5 questions, each rated on a 6-point Likert scale from 0 (not present) to 5 (constantly present). Total raw score was transformed into a percentage score ranging from 0 (worst possible quality of life) to 100 (best possible quality of life).
Time Frame: Baseline, Week 26
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 484 | 476
scores on a scale | -1.16 (0.751) | 0.22 (0.758)

9. Secondary Outcome: Percentage of Participants Requiring Rescue Therapy Over the 26 Weeks of Treatment
Description: Routine fasting self-monitored plasma glucose (SMPG) and central laboratory FPG (and HbA1c after Week 14) values were used to determine the requirement of rescue medication. Threshold values at Week 14: FPG >200 mg/dL (11 mmol/L), or HbA1c >8.5%.
Time Frame: Baseline up to Week 26
Population: ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 506
percentage of participants | 3.7 | 2.6

10. Other Pre Specified Outcome: Percentage of Participants With Hypoglycemia (Any Hypoglycemia, Documented Symptomatic Hypoglycemia, Severe and/or Confirmed Hypoglycemia) During the 26 Weeks of Treatment
Description: Hypoglycemia events were hypoglycemia of any category, severe hypoglycemia (an event that required assistance of another person to actively administer carbohydrate, glucagon, or other resuscitative actions); documented symptomatic hypoglycemia (symptoms of hypoglycemia with plasma glucose ≤3.9 mmol/L [70 mg/dL]); confirmed hypoglycemia (with or without symptoms of hypoglycemia and plasma glucose ≤3.9 mmol/L).
Time Frame: Baseline up to Week 26
Population: Safety population included all randomized participants who actually received at least 1 dose or part of a dose of investigational medicinal product (IMP) and analyzed according to the treatment actually received.
Measure: Number; unit: percentage of participants
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 505
percentage of participants
  Any hypoglycemia | 62.6 | 66.5
  Documented symptomatic hypoglycemia | 32.9 | 34.7
  Severe and/or confirmed hypoglycemia | 58.1 | 60.6
  Severe and/or confirmed hypoglycemia:<75 years age: number analyzed (Participants) | 373 | 399
  Severe and/or confirmed hypoglycemia:<75 years age | 59.2 | 60.9
  Severe and/or confirmed hypoglycemia:≥75 years age: number analyzed (Participants) | 135 | 106
  Severe and/or confirmed hypoglycemia:≥75 years age | 54.8 | 59.4

11. Other Pre Specified Outcome: Hypoglycemia (Any Hypoglycemia, Documented Symptomatic Hypoglycemia, Severe and/or Confirmed Hypoglycemia) Event Rate Per Participant Year During the 26 Weeks of Treatment
Description: as for outcome 10
Time Frame: Baseline up to Week 26
Population: Safety population.
Measure: Number; unit: events per participant year
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 505
events per participant year
  Any hypoglycemia | 6.06 | 7.74
  Documented symptomatic hypoglycemia | 1.85 | 2.56
  Severe and/or confirmed hypoglycemia | 5.17 | 6.36

12. Post Hoc Outcome: Hypoglycemia (Any Hypoglycemia, Documented Symptomatic Hypoglycemia, Severe and/or Confirmed Hypoglycemia) Event Rate Per Participant Year: By Age Categorical Data During the 26 Weeks of Treatment
Description: as for outcome 10
Time Frame: Baseline up to Week 26
Population: Safety population.
Measure: Number; unit: events per participant year
Arm/Group | HOE901-U300 | Lantus
Number analyzed (Participants) | 508 | 505
events per participant year
  Any hypoglycemia:<75 years age: number analyzed (Participants) | 373 | 399
  Any hypoglycemia:<75 years age | 6.44 | 7.85
  Any hypoglycemia:≥75 years age: number analyzed (Participants) | 135 | 106
  Any hypoglycemia:≥75 years age | 5.01 | 7.32
  Documented symptomatic hypoglycemia:<75 years age: number analyzed (Participants) | 373 | 399
  Documented symptomatic hypoglycemia:<75 years age | 2.11 | 2.52
  Documented symptomatic hypoglycemia:≥75 years age: number analyzed (Participants) | 135 | 106
  Documented symptomatic hypoglycemia:≥75 years age | 1.12 | 2.71
  Severe and/or confirmed hypoglycemia:<75 years age: number analyzed (Participants) | 373 | 399
  Severe and/or confirmed hypoglycemia:<75 years age | 5.43 | 6.37
  Severe and/or confirmed hypoglycemia:≥75 years age: number analyzed (Participants) | 135 | 106
  Severe and/or confirmed hypoglycemia:≥75 years age | 4.46 | 6.28

ADVERSE EVENTS:
Time Frame: All Adverse Events (AE) were collected from signature of the informed consent form up to the final visit (Day 184) regardless of seriousness or relationship to IMP.
Description: Reported AEs and deaths were treatment emergent that is AEs that developed/worsened and deaths that occurred during 'on treatment period' (from first dose of IMP injection up to 2 days after the last injection of IMP, regardless of introduction of rescue therapy). Analysis was performed using safety population which included all the treated participants.
Arm/Group | HOE901-U300 | Lantus
All-Cause Mortality (participants affected / at risk) | 1/508 | 0/505
Serious Adverse Events (participants affected / at risk) | 41/508 | 34/505
Other Adverse Events (participants affected / at risk) | 62/508 | 64/505
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=508) | Lantus (N=505)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute left ventricular failure (Cardiac disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 2 | 1
Angina unstable (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 2
Atrioventricular block (Cardiac disorders) | 1 | 0
Cardiac failure chronic (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 2 | 2
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Sinus node dysfunction (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Adrenal mass (Endocrine disorders) | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Arthritis infective (Infections and infestations) | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 0 | 1
Empyema (Infections and infestations) | 0 | 1
Endocarditis bacterial (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 0 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Perirectal abscess (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 3
Pyelonephritis (Infections and infestations) | 0 | 2
Urosepsis (Infections and infestations) | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Heart injury (Injury, poisoning and procedural complications) | 0 | 1
Hepatic enzyme increased (Investigations) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Chondrocalcinosis pyrophosphate (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Embolic stroke (Nervous system disorders) | 1 | 0
Hypoglycaemic coma (Nervous system disorders) | 1 | 0
Hypoglycaemic unconsciousness (Nervous system disorders) | 1 | 0
IIIrd nerve paresis (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Loss of consciousness (Nervous system disorders) | 1 | 0
Neuromyopathy (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0
Renal colic (Renal and urinary disorders) | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0
Breast mass (Reproductive system and breast disorders) | 0 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 2
Peripheral venous disease (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | HOE901-U300 (N=508) | Lantus (N=505)
Nasopharyngitis (Infections and infestations) | 37 | 38
Upper respiratory tract infection (Infections and infestations) | 27 | 28

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.